CLINICAL TRIAL: NCT04506762
Title: Does Bilateral Continuous Peri Operative Erector Spinae Plane Block Improve The Enhanced Recovery Program After Open Heart Surgeries in Adults?
Brief Title: Benefit of Peri-operative Bilateral ESP Catheters for Enhanced Recovery for Cardiac Surgery (ERCS)
Acronym: ESP_ERCS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Surgical team resigned from our hospital
Sponsor: Vinmec Healthcare System (Other)
Responsible Party: Principal Investigator, Philippe Macaire, MD, Vinmec Healthcare System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: ESP ERCS
Record Dates: First submitted 2020-08-04; First posted 2020-08-10 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Open Heart Surgery
Keywords: Erector spinae Catheter; Enhanced Recovery after Cardiac Surgery; Peri operative regional analgesia for open heart surgery; Quality of recovery

STUDY DESIGN:
Intervention Model Description: Randomized Prospective Controled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard of care for peri operative analgesia
- Intervention (Experimental): Bilateral ESP catheters for peri operative regional analgesia
  Interventions: Procedure: Regional analgesia

INTERVENTIONS:
Procedure: Regional analgesia — Insertion of bilateral ESP catheters
  Arms: Intervention

SUMMARY:
To demonstrate if the addition of peri-operative regional analgesia by Bilateral ESP catheters improves the enhanced recovery program after open heart surgeries for the duration of hospitalisation, quality of analgesia, Consumption of peri-operative opioids, quality of recovery and quality of life.

Patients will be randomly divided in 2 groups Group 1 With the actual standards of care for enhanced recovery after cardiac surgery including opioid sparing peri operative analgesia Group 2 With the actual standards of care for enhanced recovery after cardiac surgery replacing the opioid analgesia by a peri operative analgesia by bilateral ESP catheters

DETAILED DESCRIPTION:
I. CONSULTING PHASE: 1 WEEK BEFORE SURGERY

1. Preoperative information, education and counselling: patient and families receive dedicated preoperative counselling including information packets.
2. Preoperative optimization: medical optimization before surgery, including renal, pulmonary, and endocrine function.
3. Smoking and alcohol cessation: smoking and alcohol cessation advised and promoted before surgery.
4. Preoperative nutrition status: patients screened for nutritional status and counselling given for a protein-rich diet at least the week before the surgery.

II. PREOPERATIVE PHASE: 2 DAYS BEFORE SURGERY

1. Preoperative fasting and carbohydrate treatment: patients are kept NPO 8h before surgery except for oral carbohydrate beverage given 2-4h before surgery.
2. Reviewed all examination results: cardiac echography, X-ray, biology's tests
3. Consents signed.
4. Authorization operative be signed
5. Preoperative multimodal analgesic initiated : before surgery 2 h Gabapentin: 600 mg (P.O) Acetaminophen: 500 mg (P.O) Hydroxyzine: 50 mg (P.O)

III. INTRAOPERATIVE PHASE:

1. Monitoring: Usual Monitoring for Open heart surgery plus a pain monitor Ani

   •
2. Anesthesia:

   Drugs Ketamine Ketamin: 0,10 mg/kg (bolus) then 0.10 mcg/kg/h Propofol TCI mode Target Entropy from 40-60 Sufentanil 1 mcg/kg (bolus for Intubation) then 0,1-1 mcg/kg/min (50 < ANI , 70) Esmeron 0.6 - 1 mg/kg (bolus pour intubation) (TOF = 0) then 0.3 mg/kg/h 0.6 - 1 mg/kg (bolus pour intubation) (TOF = 0) then 0.3 mg/kg/h Esomeprazole 40 mg (IV) Dexamethasone 0.1 mg/kg Magnesium 10 mg/kg then 10 mg/kg/h Antibio-prophylaxy Cefazolin 2g (IV) or vancomycin 15 mg/kg before incision 1 hours.

   erector spinae plane (ESP) block insertion cathter 30 - 40 kg = 6 mL / side 40 - 50 kg = 8 mL / side 50 - 60 kg = 10 mL / side 60 - 70 kg = 12 mL / side > 70 kg = 14 mL / side

   Tramexamic Acid 2 g ( IV) 2 g (IV) Heparin 3mg/kg (bolus in Central line), 25 mg in By Pass 3mg/kg (bolus in Central line), 25 mg in By Pass

   ESP catheter Performance (Kit epidural for adult Tuohy needle 19 G Catheter 20G) It is strictly forbidden to withdraw the inserted catheter throw the needle. If you need to retrieve the catheter you must retrieve the needle with the catheter.

   Patient in Right Lateral decubitus only if Hemodynamic stable US control of needle tip (dextrose 5%) Insertion of Catheter 20G under US visualization Tip to the top of the next transverse process Test the catheter with dextrose and see the spread of the liquid under US guidance in the interfascial space anterior to the ES muscle.
   * Induction 30 min before incision
   * Identify the 2 catheters by Yellow labels (Regional analgesia code)
   * No Variation of BP during sternotomy = ESP efficient If not Sufentanil Bolus

   Coagulation test before to start By Pass ACT > 400 secondes BEFORE start by pass . Inform Surgeon (Do NOT START If NOT)
3. Cardiac by pass:

   • Cannulation Time Aortic Y cave Venous Sup and Inf or AtrioCave Connection to By Pass Air Lock Start By Pass = Volume 950-1000 ml (Ringer lactate, Gelofusine, Mannitol &t Natri bicarbonate.); Aortic clamp; Cardioplegia Type Cold: crystalloid 4-8 degree celsius (CUSTODIOL);

   Anaesthesia Action:

   Stop Ventilation disconnect ETtube/ VA Circuit only when Bypass provide a full hemodynamic CO= 2.4.BSA l/m2.min. in and out (message FULL FLOW from perfusionist)

   Maintenance anesthesia depth by ENTROPY 40-60, ANI >40 Perfusionist targets MAP 50-80 mmHg , CO = 2, 4. BSA (L/m2.min.) SVO2 > 75% Blood tests /30 mn (ABG , lactate, Hb, Glycemie, ACT with heparin reinjection )
4. Before Getting Out Of By Pass:

   * Anaesthesia Actions Ventilation
   * Restart Ventilation + Reconnect ETtube-> VA Circuit
   * Recruitment Manoeuvers low pressure Temperature and warming Cross clamp time Rhythm Monitoring Turn on the alarms De-Airing manoeuvres by surgeon & by anesthesiologist with Control by TEE. Evaluation the result of surgeon and EF before decision to use inotropes or not.
   * Removal Aortic Clamp and spontaneous defibrillation
   * Perfusion and vaso active drugs assistance SVR - MAP- CVP -CI-SVRI-SVV
   * Inotropes - Vasoconstrictors - Volemia
   * Removal Veinous Canule
5. After Bypass:

   * Test de pace-maker
   * Protamin: Slow IV protamine (dose protamine = dose heparin Total given)
   * Transamin : 2g (IV)
   * Ondansetron 4 mg (IV) - PONV prophylaxy
   * Blood tests 15 min after protamin: ABG Lactate, APTT, PT, FIBRINOGEN, Hb, Glycemia, NFS,
   * ACT to base line : 120-130 if not => More protamine
   * Blood transfusion if Hb < 10g/dL or Hct < 30%
   * Platelet transfusion if PLT< 80 000
   * Plasma fresh frozen transfusion if TP < 50%
   * Drains check.
   * Check coagulation total and blood gaz test
   * Ventilation recruitments manoeuvres

IV. POSTOPERATIVE PHASE:

1. CICU transfer:

   According to guidelines intubated ventilated patient transfer.
2. CICU:

   • Information according to guidelines Reception patient from OT

   • Identification of the 2 regional analgesia ESP catheters (Yellow Labels)

   • Drains check

   • Blood test on arrival ABG , Lactate, Hb, Glycemia, NFS, RP, ECG at arrival CICU

   • ABG, glycemie repeat every 4 hours

   • Sedation : Stable patient propofol 30-50 mg/h for 2 hours and stop when weaning criteria riched

   • Protocol for analgesia:

   all groups

   Paracetamol 1g/6h (infusion) Ketorolac 30 mg/8h Nefopam 100 mg/24h

   ESP Catheter with analgesia solution Micrel Pumps with intermittent automatic bolus (IAB) connected and started at T0

   Pump preparation and settings:

   -Patient 30 - 40 kg = 6 mL / side/6h

   -Patient 40 - 50 kg = 8 mL / side/6h
   * Patient 50 - 60 kg = 10 mL/ side/6h
   * Patient 60 - 70 kg = 12 mL/ side/6h
   * Patient > 70 kg = 14 mL / side/6h The bolus on the second catheter will be delayed by 1 hour Intermittent programmed bolus every 6h

   Rescue analgesia Morphine 50 mcg/kg/min if FLACC >3 or ANI < 40

   • Fluid management: goal directed fluid therapy (GDFT) controlled by hemodynamics monitoring (Flotrac): CI, SVV, SVRI, CVP.

   Glucose 5%: 01 ml/kg/h + electrolyte balance. Bilan import, export/ 6hours • Early extubation: (criteria weaning and extubation appendix 1)

   • Early mobilization: After extubation 4 hours, sitting in bed and moving thoracic.

   Analgeia protocle after extubation If Continuous infusion of morphine replace by Morphine PCA • Concentration Morphine : 50 mg/49 ml + Ketamine 50 mg • Loading dose: 1mg

   • PCA dose demand: 1 mg/dose

   • Lockout: 10 min

   • Continuous rate (basal): 0
   * Dose limit (hr): 6mg/hour

   Plan with daily goals for time out of bed and distance walked beginning as soon as the day of surgery.

   • Early feeding: No sonde gastric Prevention PONV Drinking clear liquids after extubation 4 hours, eating after 6 hours.

4. Criteria drain thoracic removal:

* Liquid of mediastenal drains = 0 ml/ 2h;
* No pleural effusion major;
* No pneumothorax major;
* ESP catheters removed 4h after drain removal;
* After ESP catheter removed analgesia in both group only by:

Efferalgan : 15-20 mg/kg/6h (P.O) Ibuprofen : 400 mg/8h (P.O) Gabapentin : 300 mg/6h (P.O) (5 days postop) 5. Discharge from CICU( criteria discharge appendix 1):

• VAS scores at rest and mob during hospitalization

* VAS scores at rest and mob at 1 month with return to normal activities

  6. Pain Evaluation:
* Patient Intubated scale FLACC , at rest and after pressure on sternum & drain mobilization every 6 hours
* Post extubation still drains VAS scale rest and Mob (sitting in bed moving thorax) ASAP after extubation and every 6h
* Localization of the pain VAS Sternum Back pain Drains
* After drains removed VAS rest and Mob ( sitting in bed moving thorax) and pain localization Pain (VAS rest ) just after Mediastinal drain removal if possible; Pain (VAS rest and mob every 8 h) in the ward; Pain at one month (VAS rest and mob).

  7. Discharge from hospital: (criteria discharge appendix 1)

ELIGIBILITY:
Inclusion Criteria:

* Open heart surgeries: Valvulopathies ( 1-2 valves, repair or replacement)
* Congenital heart disease (Risk Adjustment in Congenital Heart Surgery Category 1-2 ( VSD, ASD, T4F)
* NYHA II,
* Fraction ejection > 50%,
* PAPS < 50 mmHg.
* Male
* Female
* Age from 18-60 years old.
* Consent participation

Exclusion Criteria:

* Refusal participation.
* Allergy to LA
* Severe thoracic Scoliosis
* Valvulopathies association with :
* CABG
* BENTALL procedure
* Deficit mental
* Alcoholics,
* Heroine addicted
* Insufficient renal
* liver failure
* Endocarditis <1 year
* Stroke <3 months
* MI <3 months
* Bloc AV II or III with Pacemaker permanent

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2023-08-14 (Actual); Study Completion 2023-08-14 (Actual)

PRIMARY OUTCOMES:
Length of post operative stay in Hospital | 10 days
  Duration of hospitalisation

SECONDARY OUTCOMES:
Length of post operative stay in Intensive care unit | 3 days
  Duration of stay in Intensive care unit
Time to 1st mobilisation | 3 days
  1st Time to stand up out of bed
Quality of recovery | 1 month
  Quality of recovery using the scale QOR 16

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Macaire, MD, Principal Investigator — Vinmec Healthcare System
Locations (1):
- VinMec INternational hopspital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Noss C, Prusinkiewicz C, Nelson G, Patel PA, Augoustides JG, Gregory AJ. Enhanced Recovery for Cardiac Surgery. J Cardiothorac Vasc Anesth. 2018 Dec;32(6):2760-2770. doi: 10.1053/j.jvca.2018.01.045. Epub 2018 Jan 31. PMID 29503121
- [Background] Brown JK, Singh K, Dumitru R, Chan E, Kim MP. The Benefits of Enhanced Recovery After Surgery Programs and Their Application in Cardiothoracic Surgery. Methodist Debakey Cardiovasc J. 2018 Apr-Jun;14(2):77-88. doi: 10.14797/mdcj-14-2-77. PMID 29977464
- [Background] Williams JB, McConnell G, Allender JE, Woltz P, Kane K, Smith PK, Engelman DT, Bradford WT. One-year results from the first US-based enhanced recovery after cardiac surgery (ERAS Cardiac) program. J Thorac Cardiovasc Surg. 2019 May;157(5):1881-1888. doi: 10.1016/j.jtcvs.2018.10.164. Epub 2018 Dec 8. PMID 30665758
- [Background] Macaire P, Ho N, Nguyen T, Nguyen B, Vu V, Quach C, Roques V, Capdevila X. Ultrasound-Guided Continuous Thoracic Erector Spinae Plane Block Within an Enhanced Recovery Program Is Associated with Decreased Opioid Consumption and Improved Patient Postoperative Rehabilitation After Open Cardiac Surgery-A Patient-Matched, Controlled Before-and-After Study. J Cardiothorac Vasc Anesth. 2019 Jun;33(6):1659-1667. doi: 10.1053/j.jvca.2018.11.021. Epub 2018 Nov 19. PMID 30665850
- [Background] Milgrom LB, Brooks JA, Qi R, Bunnell K, Wuestfeld S, Beckman D. Pain levels experienced with activities after cardiac surgery. Am J Crit Care. 2004 Mar;13(2):116-25. PMID 15043239
- [Background] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079
- [Background] Wick EC, Grant MC, Wu CL. Postoperative Multimodal Analgesia Pain Management With Nonopioid Analgesics and Techniques: A Review. JAMA Surg. 2017 Jul 1;152(7):691-697. doi: 10.1001/jamasurg.2017.0898. PMID 28564673
- [Background] Bigeleisen PE, Goehner N. Novel approaches in pain management in cardiac surgery. Curr Opin Anaesthesiol. 2015 Feb;28(1):89-94. doi: 10.1097/ACO.0000000000000147. PMID 25500688
- [Background] Bignami E, Castella A, Allegri M. Postoperative Pain After Cardiac Surgery: An Open Issue. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):e24-e25. doi: 10.1053/j.jvca.2017.09.022. Epub 2017 Sep 20. No abstract available. PMID 29217242
- [Background] Carli F, Kehlet H, Baldini G, Steel A, McRae K, Slinger P, Hemmerling T, Salinas F, Neal JM. Evidence basis for regional anesthesia in multidisciplinary fast-track surgical care pathways. Reg Anesth Pain Med. 2011 Jan-Feb;36(1):63-72. doi: 10.1097/AAP.0b013e31820307f7. PMID 22002193
- [Background] Wong WT, Lai VK, Chee YE, Lee A. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2016 Sep 12;9(9):CD003587. doi: 10.1002/14651858.CD003587.pub3. PMID 27616189
- [Background] Zhu F, Lee A, Chee YE. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2012 Oct 17;10:CD003587. doi: 10.1002/14651858.CD003587.pub2. PMID 23076899
- [Background] Krishna SN, Chauhan S, Bhoi D, Kaushal B, Hasija S, Sangdup T, Bisoi AK. Bilateral Erector Spinae Plane Block for Acute Post-Surgical Pain in Adult Cardiac Surgical Patients: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2019 Feb;33(2):368-375. doi: 10.1053/j.jvca.2018.05.050. Epub 2018 Jun 4. PMID 30055991
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Nicholson A, Lowe MC, Parker J, Lewis SR, Alderson P, Smith AF. Systematic review and meta-analysis of enhanced recovery programmes in surgical patients. Br J Surg. 2014 Feb;101(3):172-88. doi: 10.1002/bjs.9394. PMID 24469618
- [Background] Engelman RM, Rousou JA, Flack JE 3rd, Deaton DW, Humphrey CB, Ellison LH, Allmendinger PD, Owen SG, Pekow PS. Fast-track recovery of the coronary bypass patient. Ann Thorac Surg. 1994 Dec;58(6):1742-6. doi: 10.1016/0003-4975(94)91674-8. PMID 7979747
- [Background] Myles PS, Daly DJ, Djaiani G, Lee A, Cheng DC. A systematic review of the safety and effectiveness of fast-track cardiac anesthesia. Anesthesiology. 2003 Oct;99(4):982-7. doi: 10.1097/00000542-200310000-00035. No abstract available. PMID 14508335
- [Background] Sola M, Ramm CJ, Kolarczyk LM, Teeter EG, Yeung M, Caranasos TG, Vavalle JP. Application of a Multidisciplinary Enhanced Recovery After Surgery Pathway to Improve Patient Outcomes After Transcatheter Aortic Valve Implantation. Am J Cardiol. 2016 Aug 1;118(3):418-23. doi: 10.1016/j.amjcard.2016.05.015. Epub 2016 May 14. PMID 27344271